CLINICAL TRIAL: NCT03211390
Title: Using Telemedicine to Improve Spasticity Diagnosis Rates
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, David Charles, Professor and Vice-Chairman of Neurology, Vanderbilt University Medical Center
Other Study IDs: 170703
Record Dates: First submitted 2017-07-04; First posted 2017-07-07 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Spasticity, Muscle; Muscular Diseases; Musculoskeletal Disease; Muscle Hypertonia; Muscle Spasticity; Neuromuscular Manifestations; Signs and Symptoms; Nervous System Diseases; Neurologic Manifestations
MeSH Terms: conditions — Muscle Spasticity; Muscular Diseases; Musculoskeletal Diseases; Muscle Hypertonia; Neuromuscular Manifestations; Signs and Symptoms; Nervous System Diseases; Neurologic Manifestations | interventions — Neurologic Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Neurological Examination — The subject will undergo elements of the neurological examination during which the movement disorders neurologist will look specifically for the presence of spasticity. If spasticity is found to be present during the examination, the neurologist will rate the severity of the spasticity in all affected limbs and record whether they would recommend treatment for spasticity, and if so, which treatment(s) they believe would be beneficial for the subject.
Diagnostic Test: Teleneurological Examination — A Vanderbilt neurologist will examine all consented residents using a telemedicine platform, with the assistance of a nurse at the subject's bedside. The neurologist will guide the nurse to perform elements of a physical examination to determine if a referral to a movement disorders neurologist is required for a spasticity consultation.

SUMMARY:
The purpose of this study is to test the reliability of using telemedicine so a neurologist can remotely identify residents of a long-term care facility who should be referred to a neurologist for an in-person spasticity consultation.

DETAILED DESCRIPTION:
The aim of this study is to improve spasticity (a form of muscle rigidity) diagnosis through validation of telemedicine as a tool for spasticity evaluation or referral. This study will test the reliability of using telemedicine so a neurologist can remotely identify residents of a long-term care facility who should be referred to a neurologist for an in-person spasticity consultation. The telemedicine referral tool will be tested for bedside implementation in all consenting participants residing in Tennessee State Veteran's Home, which is a long-term care facility in Murfreesboro, TN. Each of the 140 residents will receive one neurological examination and one physical examination guided by the teleneurologist. A medical record review will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of any race, aged 18 and above
* Resident of the selected long-term care facility
* The subject, or if appropriate their medical decision maker, is willing and able to provide written informed consent.

Exclusion Criteria:

* Subjects for whom participation in the study may cause medical harm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nursing home residents
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity of Teleneurology | Up to three months after consent is obtained
  A Vanderbilt neurologist will examine all consented residents for spasticity using a telemedicine platform, with the assistance of a nurse at the subject's bedside. The findings of the exam will be recorded by the research coordinator. Agreement on spasticity referral between the Vanderbilt neurologist who performed the teleneurological examination and the neurologist who performed the "gold standard" examination will be determined.

SECONDARY OUTCOMES:
Specificity of Teleneurology | Up to three months after consent is obtained
  A Vanderbilt neurologist will examine all consented residents for spasticity using a telemedicine platform, with the assistance of a nurse at the subject's bedside. The findings of the exam will be recorded by the research coordinator. Agreement on spasticity referral between the Vanderbilt neurologist who performed the teleneurological examination and the neurologist who performed the "gold standard" examination will be determined.
Spasticity Diagnosis | Up to three months after consent is obtained
  There is no biomarker for spasticity. Therefore, the diagnosis will be made on physician impression. A neurologist trained in movement disorders will examine each consented patient to determine if they have spasticity. The severity of the subject's spasticity will be documented, including the following measures: presence of fixed contractures and presence of pain on movement.

CONTACTS AND LOCATIONS:
Overall Officials: David Charles, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Tennessee State Veterans' Homes, Murfreesboro, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gracies JM. Pathophysiology of spastic paresis. II: Emergence of muscle overactivity. Muscle Nerve. 2005 May;31(5):552-71. doi: 10.1002/mus.20285. PMID 15714511
- [Background] Thompson AJ, Jarrett L, Lockley L, Marsden J, Stevenson VL. Clinical management of spasticity. J Neurol Neurosurg Psychiatry. 2005 Apr;76(4):459-63. doi: 10.1136/jnnp.2004.035972. No abstract available. PMID 15774425
- [Background] Pfister AA, Roberts AG, Taylor HM, Noel-Spaudling S, Damian MM, Charles PD. Spasticity in adults living in a developmental center. Arch Phys Med Rehabil. 2003 Dec;84(12):1808-12. doi: 10.1016/s0003-9993(03)00368-x. PMID 14669188
- [Background] Sommerfeld DK, Eek EU, Svensson AK, Holmqvist LW, von Arbin MH. Spasticity after stroke: its occurrence and association with motor impairments and activity limitations. Stroke. 2004 Jan;35(1):134-9. doi: 10.1161/01.STR.0000105386.05173.5E. Epub 2003 Dec 18. PMID 14684785
- [Background] Welmer AK, von Arbin M, Widen Holmqvist L, Sommerfeld DK. Spasticity and its association with functioning and health-related quality of life 18 months after stroke. Cerebrovasc Dis. 2006;21(4):247-53. doi: 10.1159/000091222. Epub 2006 Jan 27. PMID 16446538